CLINICAL TRIAL: NCT04825717
Title: A Randomized Controlled Trial to Examine the Efficacy of a Calorimetry Guided Nutritional Plan vs. the Recommended Daily Intake Guided Nutritional Plan in Weaning Chronically Ventilated Patients
Brief Title: Calorimetry Guided Nutrition vs. Recommended Daily Intake in Weaning Chronically Ventilated Patients: Double Blind RCT.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Reuth Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0014-18-RRH
Record Dates: First submitted 2021-03-15; First posted 2021-04-01 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Mechanical Ventilation
Keywords: Weaning; Mechanical Ventilation; Nutrition
MeSH Terms: interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: A randomized controlled double-blinded clinical trial. Intervention group: patients in this group will be administered nutrition and fluid plans prepared by the department dietitian using calorimetry-based measurements.
  Control group: The nutrition plans of patients in this group will be calculated by the department dietitian using the standard, currently accepted RDI (recommended dietary intake) formula. Nutrition will be administered according to these calculations.
  All patients included in this trial will receive a multivitamin supplement to prevent possible vitamin deficiencies.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patients and the treating physicians and nurses will be blind to patient's nutritional plan (Intervention VS Control group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in this group will be administered nutrition and fluid plans prepared by the department dietitian using calorimetry-based measurements
  Interventions: Other: Nutrition and fluid plans prepared using calorimetry-based measurements.
- Control group (No Intervention): Nutrition plans of patients in this group will be calculated by the department dietitian using the standard, currently accepted RDI (recommended dietary intake) formula.

INTERVENTIONS:
Other: Nutrition and fluid plans prepared using calorimetry-based measurements. — Nutrition and fluid plans prepared using calorimetry-based measurements.
  Arms: Intervention group

SUMMARY:
In this study, we intend to examine the effectiveness of an indirect calorimetry-guided nutrition plan, compared to the conventional, RDI-guided nutrition plan in mechanically ventilated patients, in terms of success rates of prolonged ventilation weaning, and shorter weaning time period.

Hypotheses: The rates of chronically ventilated patients weaned off invasive ventilation will increase by 15% in the intervention group, and the average weaning period in this group will be reduced by 10 ± 4 days.

Methods: A randomized controlled intervention trial that will include 200 chronically ventilated patients, admitted to the "Reuth" Rehabilitation Hospital, who meet the criteria for weaning from prolonged mechanical ventilation. Patients in the intervention group (n=100) will undergo precise calorimetric measurements using indirect calorimetry and will be administered with a nutrition plan in accordance with these measurements. Nutrition plans of patients in the control group (n=100) will be calculated and administered according to current RDI conventions (up to 24 Kcal/kg/day). In order to assure blinding, patients in the control group will undergo the same calorimetric measurements using indirect calorimetry, however, these results will not be used in any way to determine or influence the nutritional plan.

DETAILED DESCRIPTION:
Background: The number of patients in need of prolonged mechanical ventilation as means of life support is rapidly growing due to advancements in life-saving medical care for critically ill patients, an aging population, and the expanding use of aggressive surgical treatments. Both overfeeding and underfeeding are found to negatively affect the weaning process from mechanical ventilation. The caloric demands of chronically ventilated patients are reduced due to immobility and minimal energy requirements. Nowadays, nutrition plans are determined using the RDI (recommended dietary intake) formula, according to a patient's own weight and height. The RDI formula does not take into account the negligible activity levels of chronically ventilated patients or their deteriorating muscle mass, which is severely reduced due to prolonged periods of inactivity. This, in turn, may lead to increased body fat mass and fluid retention - which are both deleterious to the patients' health and may hinder their weaning from prolonged mechanical ventilation. Calorimetry is an accurate tool for measuring energy expenditures allowing us to assess the actual energy requirements of every patient. In indirect calorimetry, measurements of gas exchange are used to determine oxygen consumption versus the production and release of carbon dioxide. The "Reuth" Rehabilitation Hospital houses 108 chronically ventilated adult patients at a given moment, with turnover rates of 70-80 patients per year. If possible, these patients eventually undergo ventilation weaning. The current success rate for ventilation weaning reaches 55%, with a total duration of approximately two months.

Aim: To increase the success rates of prolonged ventilation weaning, i.e achieve a higher percentage of patients who successfully undergo mechanical ventilation weaning, with a shorter overall weaning time.

Hypotheses: The rates of chronically ventilated patients weaned off invasive ventilation will increase to 70% in the intervention group, and the average weaning period will be reduced by 10 ± 4 days.

Methods: A randomized controlled intervention trial that will include 200 chronically ventilated patients admitted to the "Reuth" Rehabilitation Hospital, who meet the criteria for weaning from prolonged mechanical ventilation. Patients in the intervention group (n=100) will undergo precise calorimetric measurements using indirect calorimetry and will be administered with a nutrition plan in accordance with these measurements. Nutrition plans of patients in the control group (n=100) will be calculated and administered according to current RDI conventions (up to 24 Kcal/kg/day). In order to assure blinding, patients in the control group will undergo the same calorimetric measurements using indirect calorimetry, however, these results will not be used in any way to determine or influence the nutritional plan.

Significance: In the United States, the use of prolonged mechanical ventilation increases by 5.5% annually, while total admissions rates increase by just 1% per year. According to estimates, the total number of patients requiring prolonged mechanical ventilation will be doubled by 2020, reaching 305,898 cases. It is safe to assume that similar trends exist in Israel, where 635 hospital beds are allocated to the ventilated patients. The total monthly admission costs for every ventilated patient in Israel are estimated at 14,140 USD, reaching nine million USD a year. Prolonged mechanical ventilation has a negative impact on both the patient and his family while caring for ventilated patients imposes a heavy burden on the health care system. In this study, we strive to increase the success rates of prolonged ventilation weaning, thereby improving ventilated patients' outcomes and alleviating the hardships inflicted on the patients, their families, and the health care system as a whole.

ELIGIBILITY:
Inclusion Criteria:

1. Newly admitted prolonged mechanical ventilation patients on tracheostomy tube ventilation (over 21 days, a minimum of 6 hours a day);
2. Over 18 years of age;
3. PEEP below 8 cm H2O;
4. FiO2 below 60%;
5. Hemodynamically stable:

   * Alert and oriented (does not apply to patients in a vegetative state);
   * Blood pressure at or above 80/50 mmHg;
   * Body temperature - normal around 36.6°C;
   * Heart rate - 40-140 beats per minute;
   * Breath - 10-20 breaths per minute;
6. No active infection (clinically stable patients receiving antibiotic treatment for more than 48 hours following an acute infection may be enrolled in the trial);

Exclusion Criteria:

1. Ventilated patients with PEEP values exceeding 8 cmH2O, which mandates the use of FiO2 values over 60%;
2. Hemodynamically unstable patients:

   * Blood pressure below 80/50 mmHg;
   * Over 140 beats per minute, or less than 40 beats per minute in symptomatic patients;
   * Newly diagnosed fever (over 38.0°C);
3. Patients receiving antibiotics for an active infection, under 48 hours.
4. Blood pH values below 7.3 due to metabolic abnormality;
5. Patients with irreversible advanced musculoskeletal neurodegenerative disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful weaning | Within 8 weeks
  Rate of successful weaning, i.e. a number of patients successfully weaned from prolonged mechanical ventilation, out of those who underwent weaning attempts.
Time to successful weaning | Within 8 weeks
  Time period in days from randomization to one of the studies groups and until successful weaning or 5 failed consecutive weaning attempts.

SECONDARY OUTCOMES:
Discharge destination following successful weaning | Within 8 weeks
  Discharge destination (other department, other hospital, home, nursing home)
Three months survival rates post-weaning | 3 months
  Three months survival rates of patients who underwent successful weaning from mechanical ventilation.

OTHER OUTCOMES:
Twelve months survival rates post-weaning | 12 months
  Twelve months survival rates of patients who underwent successful weaning from mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Reuth Rehabilitation Hospital, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fradkin M, Elyashiv M, Brik M, Kait MG, Albukrek D, Singer P, Dankner R. The efficacy of calorimetry-based nutritional support versus recommended dietary intake-based nutritional support in the successful weaning of chronically ventilated patients: A study protocol for a double blind randomized controlled trial. Clin Nutr ESPEN. 2023 Apr;54:94-97. doi: 10.1016/j.clnesp.2023.01.003. Epub 2023 Jan 13. PMID 36963903